CLINICAL TRIAL: NCT04670835
Title: Modeling the Impact of Inbound Call Distribution Virtualization in Emergency Medical Communication Centers (EMCCs) on Their Service Level
Acronym: CALL_SAMU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: IMT Mines Albi - France (https://www.imt-mines-albi.fr/) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC20_0064
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Emergency Medical Service Communication Systems, Health Care
Keywords: Emergency health service, Accessibility, Virtualization, organization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case Group (unic): 1. Group/Cohort Label :
     Users of Emergency Call Centers Users of French territory 'Region Pays de la Loire'
  2. Group/Cohort Description:
  All Users calling through the five Emergency Medical Centers of the French Pays de la Loire region (5 areas of the region are : Loire-Atlantique, Maine-et-Loire, Mayenne, Sarthe, Vendée).
  In each Emergency Medical Center, an advanced telephone system automatically keeps track of all inbound calls.
  Average annual number of incoming calls for the 5 Emergency Medical Center of Pays de la Loire region is 1,6 million.

SUMMARY:
Fast access to the Emergency Medical Communication Center (EMCC) is essential for the population in emergency situation. It is therefore essential that these call centers operate quickly and provide good quality service. However, in recent years, EMCCs have experienced a constant and increasing demand from the population. Thus, maintaining the current organization of emergency medical communication centers raises questions about both the volume of incoming calls to EMCCs and the economic constraints, which make it difficult to manage call peaks, especially in periods of crisis.

The aim of our study is to assess the impact of incoming call distribution virtualization in EMCCs on their service quality.

DETAILED DESCRIPTION:
France is facing political decisions on the evolution of Emergency Medical Communication Center organization to improve population accessibility. Regarding the performance targets requested by the French government (MARCUS report: http://www.urgences113.fr/marcus/Rapport_MARCUS3.pdf), the virtualization of inbound call distribution could improve EMCC service quality indicators.

The Virtualization is a process that consists of centralizing calls from different territories before distributing them to the centers concerned according to their availability. The objective through this process is to improve the population' access to the EMCC by reducing waits time. And on the other hand, to optimize the activity rate of dispatchers and physicians.

ELIGIBILITY:
Inclusion Criteria:

* All incoming calls passing through the five Emergency Medical Centers in the Pays de la Loire region (Loire-Atlantique, Maine-et-Loire, Mayenne, Sarthe and Vendée). In each center, an advanced telephone system automatically keeps track of all inbound calls.

Exclusion Criteria:

According to the French national consortium, incoming calls that hung up in less than 10 seconds are considered as dialing errors and are excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Users calling through the five Emergency Medical Centers of the French Pays de la Loire region (5 areas of the region are : Loire-Atlantique, Maine-et-Loire, Mayenne, Sarthe, Vendée).
  In each Emergency Medical Center, an advanced telephone system automatically keeps track of all inbound calls.
  Average annual number of incoming calls for the 5 Emergency Medical Center of Pays de la Loire region is 1,6 million.
Sampling Method: Non-Probability Sample
Enrollment: 1500000 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2021-12-16 (Estimated); Study Completion 2022-12-16 (Estimated)

PRIMARY OUTCOMES:
Operational level of service, defined by the quality of service at 20 s (QS20). It corresponds to the rate of answered calls within 20 s | 20 seconds
  This indicator is one of the most frequently used internationally to measure the performance of emergency call centers

CONTACTS AND LOCATIONS:
Overall Officials: Yann Penverne, MD, Principal Investigator — Nantes University Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Presentation of the study context; description of the protocol and his main objectives. Presentation of the team — https://www.chu-nantes.fr/recherche-clinique-26